CLINICAL TRIAL: NCT07406217
Title: OPtimisation of Antiviral Therapy in Immunocompromised COVID-19 Patients: a Randomized Factorial Controlled Strategy Trial: the SWISS OPTICOV Study
Brief Title: OPtimisation of Antiviral Therapy in Immunocompromised COVID-19 Patients: a Randomized Factorial Controlled Strategy Trial
Acronym: SWISS OPTICOV
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Calmy Alexandra (Other)
Collaborators: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor-Investigator, Calmy Alexandra, Prof, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-01720; 62987 (Other: HumRes); FNS 320003B_212963 (Other: Swiss National Fundation)
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: COVID-19; Immunodeficiency
Keywords: COVID-19; Immunodepression; SARS-CoV-2; Paxlovid; Veklury; Viral load
MeSH Terms: conditions — COVID-19; Immunologic Deficiency Syndromes | interventions — nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Nirmatrelvir/r 5 days alone (Other): Nirmatrelvir/r 300mg/100 mg bid will be given for 5 days, orally. Nirmatrelvir/r is a combination of two molecules: nirmatrelvir which is a protease inhibitor (against 3CL) and ritonavir which has a booster role. Nirmatrelvir/r (marketed by Pfizer under the brand name Paxlovid®) is indicated for the treatment of COVID-19 in adults who do not require supplemental oxygen and who are at increased risk for progressing to severe COVID-19. Paxlovid for 5 days is the standard of care.
  Interventions: Drug: Paxlovid 5 days
- Nirmatrelvir/r 10 days alone (Experimental): Intervention Nirmatrelvir/r 300mg/100 mg bid will be given for 10 days, orally.
  Interventions: Drug: Paxlovid 10 days
- Nirmatrelvir/r 5 days + remdesivir single dose (Experimental): Nirmatrelvir/r 300mg/100 mg bid will be given for 5 days, orally. Nirmatrelvir/r is a combination of two molecules: nirmatrelvir which is a protease inhibitor (against 3CL) and ritonavir which has a booster role. Nirmatrelvir/r (marketed by Pfizer under the brand name Paxlovid®) is indicated for the treatment of COVID-19 in adults who do not require supplemental oxygen and who are at increased risk for progressing to severe COVID-19. Remdesivir "flash", 200mg, intravenous. Remdesivir (marketed by Gilead under de brand name Veklury®) is indicated in patients with pneumonia requiring supplemental oxygen (inpatients), as well as in outpatients who are at increased risk of progressing to severe COVID-19. The mode of action characterize remdesivir as a direct-acting antiviral compound.
  Interventions: Drug: Paxlovid 5 days
- Nirmatrelvir/r 10 days + remdesivir single dose (Experimental): Nirmatrelvir/r 300mg/100 mg bid will be given for 10 days, orally. Remdesivir "flash", 200mg, intravenous. Remdesivir (marketed by Gilead under de brand name Veklury®) is indicated in patients with pneumonia requiring supplemental oxygen (inpatients), as well as in outpatients who are at increased risk of progressing to severe COVID-19. The mode of action characterize remdesivir as a direct-acting antiviral compound.
  Interventions: Drug: Paxlovid 10 days

INTERVENTIONS:
Drug: Paxlovid 5 days — Nirmatrelvir/r 300mg/100 mg bid will be given for 5 days, orally. Nirmatrelvir/r is a combination of two molecules: nirmatrelvir which is a protease inhibitor (against 3CL) and ritonavir which has a booster role. Nirmatrelvir/r (marketed by Pfizer under the brand name Paxlovid®) is indicated for the treatment of COVID-19 in adults who do not require supplemental oxygen and who are at increased risk for progressing to severe COVID-19.
  Arms: Nirmatrelvir/r 5 days + remdesivir single dose; Nirmatrelvir/r 5 days alone
Drug: Paxlovid 10 days — Nirmatrelvir/r 300mg/100 mg bid will be given for 10 days, orally.
  Arms: Nirmatrelvir/r 10 days + remdesivir single dose; Nirmatrelvir/r 10 days alone

SUMMARY:
The overall purpose of the trial is to evaluate the efficacy and safety of possible combination antiviral therapy direct antiviral agents (remdesivir + nirmatrelvir/r) versus the reference monotherapy (nirmatrelvir/r alone) and to assess the efficacy and safety of increasing the nirmatrelvir/r course from 5- to 10 days in immunocompromised patients diagnosed with asymptomatic or mild to moderate COVID-19.

DETAILED DESCRIPTION:
This is a randomized, controlled, factorial, superiority trial to evaluate the viral efficacy of direct antiviral agent nirmatrelvir/r + direct antiviral agent remdesivir versus nirmatrelvir/r alone and of 5 days versus 10 days of nirmatrelvir/r in immunocompromised patients diagnosed with asymptomatic or mild to moderate COVID-19. The primary objective is to assess whether (i) a combination antiviral therapy of two antiviral agents (nirmatrelvir/r + remdesivir and/or (ii) an increase in nirmatrelvir/ r duration from 5 to 10 days improves viral efficacy by decreasing the SARS-CoV- 2 positivity rate by real time RT-PCR (CT<32) in nasopharyngeal swabs at D10. Patients will be eligible if they are immunocompromised, have confirmed asymptomatic SARS-CoV-2 infection or mild to moderate COVID-19, regardless of symptoms onset, provided that they have no contra-indication to any of the study drugs. A total of 256 patients will be recruited in Switzerland and in France, Italy and Norway (through the parallel protocol ANRS0176s OPTICOV).

Participants not eligible for randomisation or who refuse to participate to the trial for any reason will be proposed to be included in an exploratory non comparative cohort (maximum 97 participants, active only in Switzerland).

ELIGIBILITY:
Inclusion Criteria:

1. Laboratory confirmed SARS-CoV-2 infection by RT-PCR or positive antigenic test (commercialized assay)
2. Asymptomatic or mild to moderate COVID-19 (WHO progression scale <5. Patients receiving oxygen therapy for reasons other than a pulmonary COVID-19 are eligible).
3. ≥ 16 years of age;
4. Immunocompromised as defined by ≥ 1 risk factors for severe COVID-19 as assessed by the FOPH list (criteria 5: diseases/treatments leading to immune suppression) or other immunosuppression criteria such as:

   * Severe immunosuppression (e.g., HIV infection with CD4 + T cell count <350 / μl)
   * Neutropenia (<1000 neutrophils / μl) ≥1 week
   * Lymphocytopenia (<200 lymphocytes/μl)
   * On dialysis treatment
   * Hereditary immunodeficiencies
   * Intake of drugs which suppress the immune system (e.g. glucocorticoids for a long time [an equivalent dose of prednisone >20 mg/day > 3 months], monoclonal antibodies, cytostatics, biological products, everolimus, mTOR inhibitors etc.) in the last 12 months
   * Active cancer under cytostatics or targeted therapy known to be immunosuppressive (e.g., platinum salts, cyclophosphamide, anthracyclines, taxanes, 5-fluorouracil, gemcitabine, purine inhibitors, proteasome inhibitors) or associated with hematologic toxicity (neutropenia, lymphopenia), for example sunitinib, imatinib, regorafenib.
   * Aggressive lymphomas (all types)
   * Acute lymphatic leukemia
   * Acute myeloid leukemia
   * Acute promyelocytic leukemia
   * T prolymphocytic leukemia
   * Primary central nervous system lymphoma
   * Stem cell transplantation
   * Light chain amyloidosis
   * Chronic lymphoid leukemia
   * Multiple myeloma
   * Sickle cell disease
   * Bone marrow transplant
   * Organ transplant
   * Being on the waiting list for an organ transplant
5. Willing and able to comply with study requirements and restrictions as described in the informed consent form (ICF)
6. Enrolled in or a beneficiary of a Social Security program (State Medical Aid (AME) is not a Social Security program) or holders of health insurance.
7. Participant's or its legal representative's signature of the informed consent form

Exclusion Criteria:

1. SARS-CoV-2 PCR ≥30 CT at screening
2. Hypersensitivity to study drugs (active substance(s) or excipients)
3. Body weight < 40 kg
4. AST and/or ALT > 5 times the upper limit
5. Cirrhosis Child-Pugh score C
6. Is taking or is anticipated to require any prohibited therapies*.
7. Participation in another interventional clinical study with an investigational compound or device, including COVID-19 therapeutics, where the study intervention is performed in the 28 days preceding the inclusion and the 10 days after the inclusion. Investigators of the different clinical studies should agree on participant's inclusion.
8. Presence of any condition for which, in the opinion of the investigator, participation would not be in participant's best interest or that could prevent, limit, or confound the protocol-specified assessments
9. Having received antiviral treatments against SARS-CoV-2 in the 14 days before the inclusion with exception of those having received one or two doses of nirmatrevir/r in the 24h preceding the inclusion in the study.
10. Pregnant or breastfeeding female

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Virological | Day 10
  Percentage of patients with SARS-CoV-2 viral load <32 CT by real-time RT-PCR in nasopharyngeal swabs at D10 after treatment initiation.

SECONDARY OUTCOMES:
Virological | Day 5, Day 14, Day 21
  Percentage of patients with SARS-CoV-2 viral load <32 CT by real-time RT-PCR in nasopharyngeal swabs at D5, D14 and D21 after treatment initiation
Virological | Day 5, Day 10, Day 14
  Percentage of patients with detectable SARS-CoV-2 viremia at D5, D10 and D14
Virological | Day 5, Day 10, Day 14, Day 21
  Decrease of SARS-CoV-2 viral load measured by copies/ml by nasopharyngeal swab at D5, D10, D14, D21 and at D5, D10 and D14 in blood samples comparatively to screening
Virological | Day 5, Day 10, Day 14, Day 21
  Number of de novo mutations after sequencing on nasopharyngeal swabs at D5, D10, D14 and D21 comparatively to screening
Virological | Day 5, Day 10, Day 14, Day 21
  To assess the phenotypic resistance (IC50 increase) against treatment for viral strains cultured from nasopharyngeal swabs at D5, D10, D14 and D21 comparatively to screening
Virological | Day 90
  Time to first negative SARS-CoV-2 RT-PCR (CT<32) until D90
Virological | Day 5, Day 10, Day 14, Day 21
  Absence of ability to cultivate virus from viral cultures from nasopharyngeal swabs at D5, D10, D14 and D21
Clinical | Day 5, Day 10, Day14, Day 21, Day 28
  Percentage of patients with sustained resolution or abatement of symptoms defined as a FLU-PRO-Plus score ≤1 at D5, D10, D14, D21 and D28
Clinical | Day 28
  All-cause hospitalization and/or death at D28
Clinical | Day 28
  Hospitalization at D28
Clinical | Day 28
  Death at D28
Clinical | Day 5, Day 10, Day 14, Day 21, Day 28, Day 90
  FLU-PRO-Plus scale at D5, D10, D14, D21, D28 and D90
Clinical | Day 90
  Rate of Post-COVID19 condition at D90 according to the WHO October 2021 definition
Clinical | Day 90
  Percentage of participants with an adverse event (AE) or serious adverse event (SAE) or AE leading to treatment discontinuation up to D90
Clinical | Day 5, Day 10
  Adherence to nirmatrelvir/r with patient-reported adherence and nirmatrelvir/r residual plasma dosage at D5 and D10, if applicable
Clinical | Day 10
  Number of drud-drug interactions who led to dosage adjustment of other patient's drugs
Clinical | Day 10
  Immunosuppressors residual concentrations, if applicable
Clinical | Day 90
  Percentage of patients with specific retreatment (by antiviral, anti-inflammatory drug or convalescent plasma) through D90
Clinical | Day 10
  Number of DDIs which led to dosage adjustment of other patient's drugs

OTHER OUTCOMES:
Safety outcome | Day 90
  Percentage of participants with an adverse event (AE) or serious adverse event (SAE) or AE leading to treatment discontinuation up to D90

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Calmy, MD PhD, Principal Investigator — Hopitaux Universitaires de Genève; Nina Khanna, MD PhD, Principal Investigator — Basel University Hospital; Nicolas Muller, MD PhD, Principal Investigator — University of Zurich; Oriol Manuel, MD PhD, Principal Investigator — University Hospital CHUV
Locations (4):
- Switzerland (4):
  - Basel University Hospital, Basel, Basel
  - Hôpitaux Universitaires de Genève, Geneva, Canton of Geneva
  - CHUV, Lausanne, Canton of Vaud
  - University Hospital Zurich, Zurich, Canton of Zurich

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data are described in the study protocol